CLINICAL TRIAL: NCT01048320
Title: A Phase I Study of Gemcitabine Plus Oxaliplatin in Combination With Imatinib Mesylate (Glivec) in Patients With Gemcitabine-refractory Advanced Adenocarcinoma of the Pancreas
Brief Title: Gemcitabine and Oxaliplatin (Gem-Ox) Plus Glivec in Gemcitabine-refractory Pancreatic Cancer
Acronym: RPGOG1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Professor David Cunningham, Royal Marsden NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR2731; EudraCT No: 2005-004022-99
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Advanced Pancreatic Cancer
Keywords: pancreatic cancer; toxicity; chemotherapy; dose finding
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other): Gemcitabine plus Oxaliplatin in combination with imatinib mesylate
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Imatinib

INTERVENTIONS:
Drug: Gemcitabine — The starting dose of gemcitabine will be 400 mg/m2 on day 1 of a two-week cycle.
  Gemcitabine is given on day 1 every two weeks according to the dose escalation schedule below:
  Dose level -1 200mg/m2 Dose level 1 400mg/m2 Dose level 2 600mg/m2 Dose level 3 800mg/m2 Dose level 4 1000mg/m2 Dose level 5 1000mg/m2 It is administered as an intravenous infusion, the lyophilized powder being diluted in normal saline, at a fixed dose of 10 mg/m2/minute.
Drug: Oxaliplatin — Oxaliplatin is given by intravenous infusion on day 2 every 2 weeks according to the dose escalation schedule below: Dose level -1 - 4 85mg/m2 Dose level 5 100mg/m2 Oxaliplatin should be diluted in 250 to 500 ml of 5% glucose solution to give a concentration not less than 0.2 mg/ml. It must be infused via a central venous line or peripheral vein over 2 hours. In the event of extravasation, administration must be discontinued immediately and the extravasation managed according to local procedures.
Drug: Imatinib — Imatinib is given for 7 days every cycle starting 2 days before the gemcitabine is given, including administration on days 1 and 2 when gemcitabine and oxaliplatin are given, and for 3 days afterwards (i.e. days -2 to +5). It is thus given on a 7 days on and 7 days off intermittent dosing schedule. The dose will be fixed at 400 mg daily in tablet form and taken once daily with food.
  Imatinib should commence either in the morning or lunchtime of day -2 and be taken at the same time daily for seven consecutive days in total.

SUMMARY:
The main research objective is to work out the optimal doses of the novel combination of gemcitabine, oxaliplatin and imatinib mesylate (glivec) in patients with advanced pancreatic cancer that has progressed during or after treatment with first-line gemcitabine.

DETAILED DESCRIPTION:
Using the phase I study design, the dose of gemcitabine will be escalated in several steps to identify the highest tolerable dose that can be given safely. Based on pre-defined dose-limiting toxicity, the maximum tolerated dose of the combination will be identified and a safer dose for further evaluation of this regimen in pancreatic cancer selected. The primary objectives are therefore based around safety of the drug combination.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* gemcitabine-refractory, histologically confirmed pancreatic cancer (progression during or within 6 months of first-line treatment)
* locally advanced or metastatic disease with measurable or non-measurable disease
* life expectancy of greater than 10 weeks
* prior treatment with investigational therapies including EGFR and VEGF antagonists is allowed when administered>4 weeks prior to start of therapy

Exclusion Criteria:

* any serious uncontrolled medical condition
* prior radiation treatment is not allowed
* no prior chemotherapy within the previous 4 weeks
* known peripheral neuropathy > CTCAE v 3.0 grade 1; absence of the deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible
* known brain metastases
* lack of physical integrity of the upper GI tract, malabsorption syndrome, or inability to take oral medication
* fertile women (<2 years after last menstruation) and men of childbearing potential not willing to use effective contraception
* pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for the study is to establish the Maximum Tolerated Dose of the drug regimen based on the endpoint of dose-limiting toxicity | 1 year

SECONDARY OUTCOMES:
Progression free survival
Overall survival
Response rate for those with measurable disease
Characterise safety profile of Gemcitabine Plus Oxaliplatin in Combination with imatinib mesylate (Glivec) in Patients with Gemcitabine-Refractory Advanced Adenocarcinoma of the Pancreas

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom